CLINICAL TRIAL: NCT05850169
Title: The Effects of Creative Dance Therapy on Motor and Executive Functions in Children With Dyslexia: A Randomized Controlled Trial
Brief Title: The Effects of Creative Dance Therapy on Motor and Executive Functions in Children With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Cemre Bafralı, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANKARAMEDİPOLUBAFRALİ002
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Dyslexia; Dance Therapy; Motor Skills; Executive Function
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): After completion of the initial assessments, the intervention group received 3 sessions per week of creative dance training for 4 weeks (12 sessions), with each session lasting approximately 40 minutes. The creative dance training took place in a 40-square-metre mirrored hall with a tatami mat on the floor. The training was conducted individually for each child in the IG. Different children's songs were selected for each session in harmony with the rhythm of the dance movements. In each session, 10 minutes of warm-up movements and 20 minutes of creative dance training were conducted, accompanied by songs. Meanwhile, materials such as spiky and heavy balls, ribbons, rhythm sticks and holihop were included in the application.
  The creative dance training was planned by diversifying the 8 movement models (breath, tactile, core-distal, head-tail, upper-lower, body side, cross lateral and vestibular) of "Brain Dance", which is a part of creative dance (Gilbert, 2002,2015).
  Interventions: Other: Creative Dance Therapy
- Control group (No Intervention)

INTERVENTIONS:
Other: Creative Dance Therapy — After completion of the initial assessments, the intervention group received 3 sessions per week of creative dance training for 4 weeks (12 sessions), with each session lasting approximately 40 minutes. The creative dance training took place in a 40-square-metre mirrored hall with a tatami mat on the floor. The training was conducted individually for each child in the IG. Different children's songs were selected for each session in harmony with the rhythm of the dance movements. In each session, 10 minutes of warm-up movements and 20 minutes of creative dance training were conducted, accompanied by songs. Meanwhile, materials such as spiky and heavy balls, ribbons, rhythm sticks and holihop were included in the application.
  The creative dance training was planned by diversifying the 8 movement models (breath, tactile, core-distal, head-tail, upper-lower, body side, cross lateral and vestibular) of "Brain Dance", which is a part of creative dance (Gilbert, 2002,2015).
  Arms: intervention group

SUMMARY:
Although some benefits of dance have been described for motor and cognitive skills, the effects on individuals with dyslexia are unclear. The purpose of this study was to investigate the effects of creative dance training on the motor and executive skills of children with dyslexia.

DETAILED DESCRIPTION:
Although some benefits of dance have been described for motor and cognitive skills, the effects on individuals with dyslexia are unclear. The purpose of this study was to investigate the effects of creative dance training on the motor and executive skills of children with dyslexia.

The randomized controlled trial was conducted between August 2019 and December 2020 in the Occupational Therapy Department of Hacettepe University. The sample consisted of 51 children with dyslexia aged 8-10 years. While 26 of the participants received routine literacy training, the other 25 also received creative dance training three times a week for 4 weeks. Motor functions were assessed using the "Bruininks-Oseretsky Motor Competence 2 Test- Short Form", and executive functions were assessedusing the "Executive Function and Occupational Routines Scale".

ELIGIBILITY:
Inclusion Criteria:

* an age between 6 and 10 years
* a diagnosis of dyslexia according to DSM-V criteria
* continued formal education in elementary school
* participation in routine literacy training in a special education and rehabilitation center
* voluntary participation in the study.

Exclusion Criteria:

* having additional physical or psychological problem accompanying the dyslexia
* using of psychotic drugs
* participating in sports regularly.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2019-08-24 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency Second Edition Brief Form, (BOT-2 SF) | 20 minutes
  Bruininks-Oseretsky Test of Motor Proficiency Second Edition Brief Form, (BOT-2 SF) was used to assess the motor functions of the participants. BOT2- SF consists of eight subdomains, including fine motor precision, fine motor integration, manual dexterity, bilateral coordination, balance, upper limb coordination, strength, speed and agility, and includes a total of 12 items (Bruininks, 2010). The test takes 15-20 minutes to complete. The higher score obtained from the test indicates a better performance in motor competence, and the highest score that can be obtained from the test is 72 points (Bruininks, 2010). The Turkish validity and reliability study of the BOT2-SF was conducted by Köse et al. (2018) on children with specific learning difficulties.
Executive Function and Occupational Routines Scale (EFORTS) | 20 minutes
  Executive Function and Occupational Routines Scale (EFORTS) was used to assess participants' executive functions. EFORTS is a 30-item scale that measures the child's daily routine and consists of three factors: morning and evening routines, play and leisure routines, and social routine (Frisch & Rosenblum, 2014). It is completed by the family and rated on a 1-5 Likert scale. A high score on each item indicates that the child performs better in an occupation that requires executive functions. The Turkish validity and reliability study was conducted by Akyürek and Bumin (2017).

CONTACTS AND LOCATIONS:
Overall Officials: Cemre Bafralı, Msc, Principal Investigator — Ankara Medipol University
Locations (1):
- Cemre Bafralı, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes